CLINICAL TRIAL: NCT02346773
Title: Effects of Omega-3 Fatty Acids Supplementation on Brain and Behaviour in Healthy Children.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Nottingham (Other)
Collaborators: Unilever R&D (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple
Other Study IDs: UNottingham
Record Dates: First submitted 2014-12-22; First posted 2015-01-27 (Estimated); Last update posted 2015-12-09 (Estimated); Status verified 2015-12

CONDITIONS: Behaviour
MeSH Terms: conditions — Behavior

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- ω-3 LC-PUFA group (Active Comparator): The intervention product was a full fat (80%) margarine. The active intervention product contained 590 mg docosahexaenoic acid (DHA) and 650 mg eicosapentaenoic acid (EPA) per 10-g daily serving.
  Interventions: Dietary Supplement: ω-3 LC-PUFA
- Placebo group (Placebo Comparator): The placebo product was a similar margarine with the same sensory properties, but with monounsaturated fatty acids (MUFA; refined plant oils) replacing EPA and DHA; total saturated fatty acids (SAFA) and ω-6 long chain polyunsaturated fatty acids (LC-PUFA) content were similar between the active and placebo products.
  Interventions: Other: Placebo

INTERVENTIONS:
Dietary Supplement: ω-3 LC-PUFA — The intervention product was a full fat (80%) margarine.Participants were provided with one-month supply of the intervention product (including reserve products) at the onset of the intervention and received a new supply monthly. The intervention products were provided in neutral serving-sized cups, each containing 10 grams of margarine.The child's parents were instructed to have their child consume one complete portion pack (10 g) of margarine per day. The margarine had to be consumed as spread on sandwiches, crackers or bread rolls.The intervention product could be consumed on various periods over the day or all at one occasion. Every day a new portion pack had to be used, even if there was margarine left in the package of the previous day.
  Arms: ω-3 LC-PUFA group
Other: Placebo — The placebo product was a similar margarine with the same sensory properties, but with monounsaturated fatty acids (MUFA; refined plant oils) replacing EPA and DHA; total saturated fatty acids (SAFA) and ω-6 long chain polyunsaturated fatty acids (LC-PUFA) content were similar between the active and placebo products.
  Arms: Placebo group

SUMMARY:
Currently, there is considerable interest in the possibility that dietary supplementation with fatty acids, mostly omega-3 fatty acids, will have potential benefits for brain development. Epidemiological and clinical studies support the idea that relative disappearance of omega-3 diet from the diet in developed countries has been linked with increases in both physical and mental disorders. Omega-3 deficiency may lead to cognitive impairment, motor dysfunction and visual acuity problems. It is further known that families with lower socioeconomic status may have poorer diet and, consequently, may not realize their full potential regarding their cognitive abilities. The aim of this project is to evaluate effectiveness of a diet intervention rich in omega-3 acid in healthy children 9-to-12 years old from less well-off families.

DETAILED DESCRIPTION:
Background It has been established that a safe environment, adequate stimulation, and parental care play a major role in brain development. An adequate diet is also critically important for brain development in growing children. It has been suggested that omega-3 fatty acids are essential to human health as well as cognitive development. Omega-3 acid is important during prenatal human brain development, especially for synaptogenesis. Levels of omega-3 amino acids in during prenatal and early postnatal (breastfeeding) periods depend on their levels in maternal circulation. Later on, omega-3 must be present in the child's diet. It seems that omega-3 deficiency may associated with impaired visual acuity, cognition, cerebellar dysfunction and other neurological disorders (Haag, 2003; Review). Thus, omega-3 supplementation may be beneficial in children with poor diet, often associated with a lower socioeconomic level (Northstone et al. 2008).

Aims and Design We assessed effects of Omega-3 supplementation on brain and behaviour of 40 healthy children 9-to-12 years old. Since diet supplementation may be beneficial in particular to children with poor diet, we recruited children in less well-off neighbourhoods, as determined by the Index of Multiple Deprivation 2007. Our aim was to examine differences on cognitive performance pre and post diet supplementation.

The brain structure was assessed using magnetic resonance imaging (MRI). Cognitive abilities as well as behavioural problems were assessed using a comprehensive battery of tests and questionnaires. To evaluate the effectiveness of the supplementation, we collected a blood sample to investigate the fatty acids level in the blood. The above assessments were carried out twice: before and after a 3-month dietary intervention.

The dietary intervention included a daily use, for a period of three months, of margarine enriched (Experimental group) or not (placebo group) with Omega-3 fatty acids. We hypothesized that this intervention will improve some cognitive deficits (such as attention, processing speed) and behavioural symptoms (e.g. depression, aggressiveness, impulsivity) together with an impact on brain structure (e.g. white-matter properties related to myelination).

Experimental Protocol Each participant participated in two phases: a clinical assessment phase (to assure exclusion and inclusion criteria) and an experimental phase. The experimental phase consisted of the baseline (pre-intervention) assessment, the diet intervention (3 months) and the post-intervention assessment.

At baseline, both groups (enriched diet and placebo) underwent a cognitive assessment and MRI. Parents were asked to complete a questionnaire about the child's behaviour and some demographical data such as number of children, education etc. Children were also asked to provide a blood sample, which was taken by a fully trained and licensed team member.

After the baseline assessment, experimental group (n=20) and control group (n=20) followed a diet supplementation with omega-3 fatty acids or placebo diet respectively. The intervention lasted for three months and then the tests were re-administered for both groups (cases and controls). Parents were also asked to complete a brief questionnaire to measure children's behaviour.

ELIGIBILITY:
Inclusion Criteria:

* Child in target age (9-12 yrs)
* Child native language English
* Child is available for providing a blood sample
* Child is available for MRI scan

Exclusion Criteria:

* 1) eating fatty fish/shellfish more than once a week;
* 2) using ω-3 and/or ω-6 LC-PUFA supplements more than once a week;
* 3) consuming products fortified with ω-3 LC-PUFA (EPA and/or DHA >100 mg/day) in the three months prior to study participation;
* 4) positive history of alcohol abuse during pregnancy;
* 5) positive history of malignancy and heart disease requiring heart surgery;
* 6) Premature birth (< 35 weeks) and/or detached placenta
* 7) Hyperbilirubinemia requiring transfusion
* 8) severe mental illness (e.g. autism, schizophrenia) or mental retardation;
* 9) MRI contraindications
* 10) Type 1 diabetes
* 11) Epilepsy
* 12) Brain tumour
* 13) Head trauma with loss of consciousness >30 minutes
* 14) Muscular dystrophy, myotonic dystrophy
* 15) Nutritional and metabolic diseases (e.g. failure to thrive, phenylketonuria)
* 16) Hearing deficit (requiring hearing aid)

Ages: 9 Years to 12 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 40 (Actual)
Dates: Start 2008-11; Primary Completion 2009-12 (Actual); Study Completion 2009-12 (Actual)

PRIMARY OUTCOMES:
Multi-modal Magnetic Resonance Imaging (MRI): Investigating the effects of three months of EPA&DHA supplementation on brain structure of healthy children 9-to-12 years old. | Change from baseline MRI measures (DTI, MTR, MRS) at 3 months

SECONDARY OUTCOMES:
Cognitive assessment as measured by neuropsychological testing | Change from baseline cognitive assessment at 3 months
  Neuropsychological testing: Intelligence Quotient (WISC-IV), Processing Speed (Trail Making Test), Selective & Sustained Attention (Ruff 2&7 Test), Working Memory (Self Ordered Pointing Test), Wisconsin Card Sorting Test

CONTACTS AND LOCATIONS:
Overall Officials: Tomáš Paus, M.D., Ph.D., Principal Investigator — Rotman Research Institute, University of Toronto, Toronto, Canada
Locations (1):
- Brain and Body Centre, School of Psychology, University of Nottingham, Nottingham, United Kingdom